CLINICAL TRIAL: NCT03269006
Title: Improved Visceral Leishmaniasis (VL) Case Detection and Vector Control to Support the VL Elimination Initiative in Bangladesh
Brief Title: Improved Case Detection and Vector Control for Visceral Leishmaniasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PR-14087
Record Dates: First submitted 2017-03-27; First posted 2017-08-31 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2019-12

CONDITIONS: Visceral Leishmaniasis
Keywords: Visceral leishmaniasis; Vector control; Sand fly,; Bangladesh
MeSH Terms: conditions — Leishmaniasis, Visceral

STUDY DESIGN:
Intervention Model Description: A randomized control trial will be performed with Inesfly 5AIGRNG TM, commercial available durable wall lining (DWL), impregnated of existing bed-net with insecticide tablet, KO TAB 123, indoor residual spraying (IRS) with Delthamethrin vs a control group (study with 5 arms). The study will be carried out in villages located in Mymensingh District. Four high endemic villages will be selected for the study. As per sample size calculation we need minimum 31 households to see the efficacy of the interventions. We will include 50 households for each intervention and 50 for control (No intervention). 18 households from each cluster will be selected randomly for entomological analysis which includes sand fly density measurement at base line and 1, 3, 6, 9, 12, 15, 18, 21 and 24 months after intervention, and WHO Cone bio-assay on the intervention surfaces and the control surfaces at 1, 3, 6, 9, 12, 15, 18, 21 and 24 months after intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Inesfly Paint (Experimental): Inesfly 5AIGRNG TM containing Alphacypermethrin 0.7%; D-Allethin 1.0% and Pyriproxyphen (0.063%). The formulation is vinyl paint with an aqueous base, with the active ingredients residing within Ca CO3 and resin microcapsules, allowing a gradual release of active ingredients. Microcapsules range from one to several hundred micrometers in size.
  Interventions: Device: Inesfly Paint
- IDWL (1m) (Experimental): Install durable wall lining up to one meter from the floor of the intervention room containing deltamethrin to kill immature stage and as well as adult sand flies.
  Interventions: Device: IDWL (1m)
- ITN (KO-Tab 123) (Experimental): impregnation of existing bed net by the insecticide tablet, K-O Tab 1-2-3 containing deltamethrin.
  Interventions: Device: ITN (KO-Tab 123)
- IRS (Delthamethrin) (Experimental): indoor residual spraying with Delthamethrin in the living rooms
  Interventions: Device: IRS (Delthamethrin)
- Control (No Intervention): without any study interventions

INTERVENTIONS:
Device: Inesfly Paint — Inesfly 5AIGRNG TM paint contain Alphacypermethrin 0.7%; D-Allethin 1.0% and Pyriproxyphen (0.063%).
  Others intervention such as IRS, ITN and IDWLcontain Delthamethrin
  Arms: Inesfly Paint
Device: IDWL (1m) — Install durable wall lining up to one meter from the floor of the intervention room containing deltamethrin to kill immature stage and as well as adult sand flies
  Arms: IDWL (1m)
Device: ITN (KO-Tab 123) — Impregnation of existing bed net by the insecticide tablet, K-O Tab 1-2-3 containing deltamethrin
  Arms: ITN (KO-Tab 123)
Device: IRS (Delthamethrin) — Indoor residual spraying with Delthamethrin in the living rooms
  Arms: IRS (Delthamethrin)

SUMMARY:
Visceral leishmaniasis (VL) also known as kala-azar is a public health problem in Bangladesh. Since 2005 a national kala-azar elimination program is going on in the country. The program has preparatory, attack, consolidation and maintenance phases. The target of the program is to reduce the VL incidence less than 1 per 10,000 people at upazila (sub-district) level in VL endemic upazilas of the country. The program is heading successfully to its consolidation phase.

During attack phase house to house search for VL suspects and also suspects with Post-kala-azar Dermal Leishmaniasis (PKDL) was the tool for early diagnosis of VL and PKDL cases. Indoor residual spraying with insecticide (Deltamethrin) was the method for sand fly control to reduce the transmission of the disease. Since in the consolidation phase the VL case load is many times less than that in the attack phase, house to house search for VL and PKDL cases and IRS for vector control is no more cost-effective for the program. Therefore there is a need for alternative methods for active search of VL and PKDL cases and method for sand fly control, appropriate for the consolidation phase.

In the present study the investigators propose to investigate the efficacy of Inesfly 5AIGRNG TM containing Alphacypermethrin 0.7%; D-Allethin 1.0% and Pyriproxyphen (0.063%), commercial available durable wall lining (DWL), impregnated of existing bed-net with insecticide tablet, KO TAB 123, indoor residual spraying (IRS) with Delthamethrin against a control group Methods: A cluster randomized controlled design to measure sand fly density reduction at intervention household as well as sand fly mortality by entomological methods.

Outcome measures/variables: reduction of sand fly density at intervention household and sand fly corrected mortality on intervention surfaces compare to control households/conditions.

DETAILED DESCRIPTION:
The objective of this study is to test the efficacy Inesfly 5AIGRNG TM containing Alphacypermethrin 0.7%; D-Allethin 1.0% and Pyriproxyphen (0.063%), and other intervention with control group. The formulation is vinyl paint with an aqueous base, with the active ingredients residing within Ca CO3 and resin microcapsules, allowing a gradual release of active ingredients. Microcapsules range from one to several hundred micrometers in size. Inesfly has been tested for control of malaria and chagas disease vector with encouraging results. The product is effective even against vectors, resistant to pyrethroids.

A randomized control trial will be performed with Inesfly 5AIGRNG TM containing Alphacypermethrin 0.7%; D-Allethin 1.0% and Pyriproxyphen (0.063%), commercial available durable wall lining (DWL), impregnated of existing bed-net with insecticide tablet, KO TAB 123, indoor residual spraying (IRS) with Delthamethrin against a control group (study with 5 arms). The study will be carried out in villages located in Mymensingh District , one of the high VL endemic district in Bangladesh. The VL burden of the villages will be estimated using the VL case reports in the last 12 months. Four high endemic villages will be selected for the study. As per sample size calculation the investigators need minimum 31 households to see the efficacy of the interventions (see sample size calculation part below). The investigators will include 50 households for each intervention and 50 for control (No intervention). Twenty-five households (HHs) from each village will be selected randomly which will be considered as a cluster. Field Research Assistant will be listed all the study households. Only subjects who agree to participate and freely signed the consent form will be included in the study. Household roster and household head interview for socio-demographic, socio-economic and knowledge about VL and VL vectors will be done. Based on sample size calculation, 18 HHs from each cluster will be selected randomly for entomological analysis which includes sand fly density measurement (base line and 1, 3, 6, 9,12, 15, 18, 21 and 24 months after intervention), WHO Cone bioassay on the intervention surfaces and control surfaces at 1, 3, 6, 9,12, 15, 18, 21 and 24 months after intervention After performing baseline sand fly density measurements, clusters will be redefined with High density (sand fly density =>50th percentile), and low (sand fly density (<50th percentile). One cluster will be selected randomly from each density group for the intervention with Inesfly, commercial DWL, and the control group with no intervention. All groups will receive the routine vector control services by the national program. Acceptability survey of the intervention will be conducted at 6 weeks since intervention to see the community acceptance of the intervention.

Entomological methods:

Sand fly collection and density measurement For the entomological activities for objective 2 and objective 3 HH head will be informed and his/her informed, written voluntary consent will be obtained before the start of any activities. HH head and members will be requested one day before by the research team to make space for conduct installation of DWL / wall paining with Inesfly by removing materials including furniture to a safe place. They also will be informed that for entomological activities i.e. for collection of sand fly by CDC light trap research team will visit the HH for two consecutive days as on day one they will visit in the evening to place CDC light trap in a corner of the main room and to take it out on the following morning. As sand fly collection will be done before intervention and at 1 month, 6 months and 12 months after intervention research team will visit the HH 4 times for sand fly collection. In addition to conduct the WHO Cone bioassay test which will be done again at 1 month, 3 months and 12 months since intervention the HH will be visited again 3 times by the research team.

Sand flies will be collected on two consecutive nights with CDC light traps by trained personnel with guidance from a member of the study team. Light traps will be kept in a corner from 6 pm to 6 am, 2 inch away from the wall with a distance of 6 inches between the floor and the bottom of the sac. The sand fly density will be expressed as number of P. argentipes per light trap per night. Sand fly identification will be done as follows:

* Upon collection, sand flies will be segregated and labeled by batch indicating the date and the pre-printed batch numbers. Sand fly numbers and sex will be identified under microscope.
* Morphological identification will be done in the field using the following criteria:

vi. Phlebotomus argentipes Pa: Black thorax+silvering shining of the tarsal tip of the leg+3mm.

vii. Phlebotomus papatasi Pp: Brown to yellow thorax+3mm. viii. Sergentomyia sp Sr:I1-2mm c. Sex and physiological status ix. Males: external genitalia with claspers x. Females: without claspers, Blood-fed, unfed, gravid (no undigested blood).

WHO Cone Bioassay Test The WHO cone bioassays will be performed using the cone method (WHOPES 2005.11) on treated and non-treated bed-nets with wild caught (manually collected) sandflies at 1 month, 6 months and 12 months after intervention. Bioassays will be carried out at room temperature at 25o- 29oC and 75-85% humidity. Resting sandflies will be collected manually by aspirator during early morning and evening. In each net, 10-12 female sand flies will be introduced in each of the cones placed against the DWL / Wall for 30 minutes. The sand flies will be then transferred from each cone to a paper cup for observation. They will be observed over 24 hours to calculate the mortality. The mortality rates of sand flies will be corrected with Abbot's formula (WHOPES 2005.11).

Measurement of efficacy of interventions: Efficacy will be defined by the reduction of sandfly density by intervention compared to control measured by sandfly density at 1 months, 6 months and 12 months after intervention; percentage mortality of sand-fly assessed by WHO Cone Bioassay test on DWL and wall after 1 months, 6 months and 12 months following intervention.

ELIGIBILITY:
Inclusion Criteria:

* Filed Research Assistant will be listed all the study households in the selected study areas.
* Only subjects who agree to participate and freely signed the consent form will be included in the study.

Exclusion Criteria:

- Subjects who will not agree to participate and freely signed the consent form will be included in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-04-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Reduction of Vector density (CDC light trap) | at base line and 1,3, 6, 9, 12, 15, 18, 21 and 24 months after intervention
  Based on sample size calculation, 18 households from each cluster will be selected randomly for sand fly density measurement at base line and 1,3, 6, 9, 12, 15, 18, 21 and 24 months after intervention

SECONDARY OUTCOMES:
Corrected sand fly mortality | at 1,3, 6, 9, 12, 15, 18, 21 and 24 months after intervention
  WHO Cone bio-assay will be done on the intervention surfaces and the control surfaces (at 18 households from each cluster) at 1, 3, 6, 9, 12, 15, 18, 21 and 24 months after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Dinesh Mondal, PhD, Principal Investigator — Senior Scientist
Locations (1):
- Icddr,B Field Site, Mymensingh, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
As per institutional (icddr,b) data sharing policy.
Supporting Information: CSR
Time Frame: As per institutional (icddr,b) data sharing policy.
Access Criteria: As per institutional (icddr,b) data sharing policy.
URL: http://www.icddrb.org/component/content/article/10003-data-policies/1893-data-policies